CLINICAL TRIAL: NCT01078870
Title: A Double-blind, Randomized, Placebo Controlled Clinical Trial on Comparing Escitalopram and Duloxetine add-on for Negative Symptoms in Schizophrenic Subjects With Neuregulin-1 (NRG1) Risk Genotype
Brief Title: Trial for Antidepressant Treatment for Negative Symptom of Schizophrenia With NRG1 Risk Genotype
Acronym: TANESN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Chih-Min Liu/M.D., National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 200907058M
Record Dates: First submitted 2010-02-28; First posted 2010-03-02 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2010-02

CONDITIONS: Schizophrenia
Keywords: Negative symptom
MeSH Terms: conditions — Schizophrenia | interventions — Escitalopram; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental)
  Interventions: Drug: Lexapro
- B (Experimental)
  Interventions: Drug: Cymbalta
- C (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lexapro — 10mg/cap 1~2# QD
  Arms: A
Drug: Cymbalta — 30mg/cap 30~60mg/QD
  Arms: B
Drug: Placebo — 1~2#/cap QD
  Arms: C

SUMMARY:
The project is a double-blind, randomized, placebo controlled clinical trial comparing 3 groups of schizophrenic subjects, who have no less than moderate degree of negative symptoms and carry the homozygous risk genotype (TT) of NRG1-P3, each group having 30 individuals, treated by add-on with escitalopram 10-20 mg/day, duloxetine 30-60 mg/day, and placebo. The treatment duration is 8 week. The investigators will evaluate the Positive and Negative Symptom Scale (PANSS) at baseline, Day 14, Day 28, Day 42, and Day 56. The primary outcome of interest will be the differences of averaged reduction of negative symptom scores among 3 groups and an average decrease of 2 or more in the negative symptoms will be indicated as improvement.

DETAILED DESCRIPTION:
Negative symptoms of schizophrenia are enduring and detrimental. The underlying pathophysiology of negative symptoms is yet to be understood. Previous clinical trials of antidepressants as add-on therapy for negative symptoms in schizophrenia patients usually found merely a trend favoring augmentation strategy. Since schizophrenia is a heterogeneous disorder, clinical studies are often unable to reveal conclusive results. Thus efforts have been made to classify relatively homogeneous groups of patients by different approaches. Here, we proposed a translational study originating from our novel results of animal study and genetic study describe as the follows.We studied the neurobiological difference of the mice with the heterozygous deletion of NRG1(NRG1+/-mice)in comparison with their wild-type littermates. It was found that the antidepressant effect of desipramine for the immobilization was markedly increased in NRG1+/-mice assessed by two models, forced swimming test and tail suspension test. Furthermore, the expression of serotonin transporter (SERT) was up-regulated in most brain regions in NRG1+/-mice, indicating that the basal activity of serotonin was reduced because of higher uptake rate in NRG1+/-mice. Our data indicate that serotonin hypo-function may be involved in the immobilization symptom of schizophrenia with NRG1 defect. Increased immobility of forced swimming test in mice was suggested to be an animal model of negative symptoms. Thus our study implied that serotonin transporter blockers may be beneficial for the treatment of negative symptoms in some subtypes of schizophrenia, especially for the patients with NRG1 defect, which could be tested by examining specific polymorphism of NRG1 gene.We have identified a novel promoter variant (TC), named NRG1-P3, located on the promoter region of type V NRG1, from a direct sequencing study in Taiwanese schizophrenic patients and found it was significantly associated with schizophrenia in a large case-control sample. Through the luciferase reporter assay, we found the promoter construct with the risk genetic variant (T allele) of NRG1-P3 has significant lower luciferase reporter activity than that with the protected allele (C allele). It implied the schizophrenic patients with the T allele of NRG1-P3 might have lower NRG1 expression than those with the C allele. It is hypothesized that the negative symptoms of the schizophrenic patients with the T allele of NRG1-P3 will be more responsive to the SSRI or SNRI treatment.The project is a double-blind, randomized, placebo controlled clinical trial comparing 3 groups of schizophrenic subjects, who have no less than moderate degree of negative symptoms and carry the homozygous risk genotype (TT) of NRG1-P3, each group having 30 individuals, treated by add-on with escitalopram 10-20 mg/day, duloxetine 30-60 mg/day, and placebo. The treatment duration is 8 week. We will evaluate the Positive and Negative Symptom Scale (PANSS) at baseline, Day 14, Day 28, Day 42, and Day 56. The primary outcome of interest will be the differences of averaged reduction of negative symptom scores among 3 groups and an average decrease of 2 or more in the negative symptoms will be indicated as improvement.The project is novel and feasible because (1) it is the first clinical trial for the treatment of negative symptoms according to different genotypes of the patients and helps fulfill the prospect of individualized medication. (2) the research findings the translational study based upon are novel and unique and comes from our research team. (3) our research team mastered in clinical studies and has many clinical resources to recruit enough patients.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 18-65
2. meet the diagnostic criteria of Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) schizophrenia
3. the genotype of NRG1-P3 is the homozygous risk genotype (TT)
4. under second-generation antipsychotic treatment with relatively stable clinical status (no change of prescribed medications during past 8 weeks and all symptom items in the positive subscale of PANSS with score no more than 4)
5. having moderate to marked negative symptoms (scores between 4 to 6 in the items of N2, emotional withdrawal, and N4, passivity/apathetic social withdrawal)

Exclusion Criteria:

1. lifetime diagnosis of schizoaffective disorder, bipolar affective disorder, and major depressive disorder and the score of Hamilton Depression Rating Scale (HAM-D) is above 18
2. the genotype of NRG1-P3 is TC or CC
3. having any major systemic illness
4. receiving first-generation antipsychotics or already on antidepressants or mood-stabilizing agents adjuvant
5. substance abuse in the past 6 months
6. pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-01 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome of interest will be the differences of averaged reduction of negative symptom scores among 3 groups compared by Analysis of Variance (ANOVA). | 2010/12

SECONDARY OUTCOMES:
A decrease of 2 or more in the items of N2 or N4 will be indicated as improvement, and the proportion of subjects meeting this improvement criterion will also be compared among three groups by Chi-square statistics | 2010/12

CONTACTS AND LOCATIONS:
Overall Officials: Liu Chih-Min, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan